CLINICAL TRIAL: NCT03145402
Title: The Effect of Intracoronary Autologous Bone Marrow Derived Mononuclear Stem Cell Transplantation in Heart Failure (HF) Patients
Brief Title: ICMNC-HF. IntraCoronary Bone Marrow MonoNuclear Cells in Heart Failure (HF) Patients
Acronym: ICMNC-HF
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SCARM Institute, Tabriz, Iran (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCARM-Heart-001
Record Dates: First submitted 2017-05-02; First posted 2017-05-09 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2019-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracoronary injection of stem cell (Experimental): Autologous bone marrow-derived mononuclear cells injection in patients with Heart Failure
  Interventions: Biological: Intracoronary injection of stem cell
- Placebo (Placebo Comparator): Placebo injection via coronary arteries in patients with Heart Failure
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Intracoronary injection of stem cell — Autologous bone marrow-derived mononuclear cells are obtained from 100-150ml of bone marrow aspirated under local anaesthesia from the iliac crest. Intracoronary infusion of the cells is performed in patients with Heart failure via conventional percutaneous intracoronary intervention techniques.
  Arms: Intracoronary injection of stem cell
Biological: Placebo — Injection of Placebo in patients with Heart failure via coronary arteries
  Arms: Placebo

SUMMARY:
This is a prospective, randomised double blind, controlled, parallel-group phase I and II study. Its aim is to assess that a single intracoronary infusion of autologous bone marrow-mononuclear cells is safe and effective in hear failure patients with reduced left ventricular ejection fraction(<=30%) when compared to a control group of patients undergoing best medical care.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women of any ethnic origin 18 ≤ aged≤ 65 years
2. EF≤40 (by Echocardiography) and regional wall motion abnormality
3. Not responding to standard therapies
4. the New York Heart Association (NYHA) class ≥ III
5. Myocardial infarction due to coronary artery atherosclerotic disease
6. An area of regional dysfunction, i.e., hypokinetic, akinetic, or dyskinetic (echocardiography or MRI)
7. Normal liver and renal function
8. No or controlled diabetes
9. Able to give voluntary written consent and understand the study information provided to him

Exclusion Criteria:

1. Participation in another clinical trial within 30 days prior randomisation
2. Previously received stem/progenitor cell therapy
3. Pregnant women
4. Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study or to follow the protocol
5. Cardiogenic shock requiring mechanical support
6. Congenital / valvular heart disease
7. Implantable cardioverter defibrillator (ICD) transplant
8. Platelet count <100.000/µl, or hemoglobin <8.5 g/dl
9. Impaired renal function, i.e. creatinine >2.5 mg/dl
10. Fever or diarrhea within 4 weeks prior screening
11. History of bleeding disorder within 3 months prior screening
12. Uncontrolled hypertension (systolic >180 mmHg and diastolic >120 mmHg) or Sustained ventricular arrhythmia
13. Life expectancy of less than two years from any non-cardiac cause or uncontrolled neoplastic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-10-20 (Estimated); Primary Completion 2021-08-28 (Estimated); Study Completion 2021-10-02 (Estimated)

PRIMARY OUTCOMES:
Death | 12 months
  The rate of patients mortality after transplantation
Hospitalization | 12 months
  the rate of hospitalization after transplantation

SECONDARY OUTCOMES:
Ejection fraction changes | 12 months
  Elevation of ejection fraction in patients after transplantation
6-minute walk test (6MWT) | 12 months
  Evaluation the improvement of 6MWT test after transplantation
Pro b-type natriuretic peptide (Pro-BNP) changes | 12 months
  Elevation the reduction of Pro-BNP in patients after transplantation
NYHA functional class | 12 months
  Evaluation the improvement of NYHA functional class in patients

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Aslanabadi, MD, Cardiologist, Study Director — Tabriz University of Medical Sciences; Mohammad Nouri, Ph.D, Study Chair — Head of SCARM institute; Peyman Keyhanvar, MD, Ph.D, Principal Investigator — Deputy for translational medicine of SCARM institute; Raheleh Farahzadi, Ph.D, Principal Investigator — Cardiovascular research center, Tabriz University of Medical Sciences, Tabriz, Iran; Yousef Faridvand, Ph.D, Principal Investigator — SCARM institute; Elgar Anamzadeh, MD, Cardiologist, Principal Investigator — Tabriz University of Medical Sciences
Locations (1):
- Stem Cell And Regenerative Medicine institute (SCARM), Tabriz, Iran

IPD SHARING:
Plan to Share IPD: No